CLINICAL TRIAL: NCT00503971
Title: Sequential Phase I/II Trial of Oral Vorinostat in Combination With Erlotinib in Non-small-cell Lung Cancer Patients With Mutations at Epidermal Growth Factor Receptor With Disease Progression After Erlotinib Treatment
Brief Title: Phase I/II of Oral Vorinostat Combination With Erlotinib in NSCLC Patients With EGFR Mutations With DP After Erlotinib.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spanish Lung Cancer Group (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TARZO; 2007-003646-15 (EudraCT Number)
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Vorinostat; NSCLC; EGFR; Erlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vorinostat plus erlotinib (Experimental): Vorinostat plus erlotinib
  Interventions: Drug: Vorinostat plus Erlotinib

INTERVENTIONS:
Drug: Vorinostat plus Erlotinib — Phase I:
  Dose level 1: 300 mg V d1-7 every 21 days plus 100 mg E daily Dose level 2: 400 mg V d1-7 every 21 days plus 100 mg E daily Dose level 2b: 300 mg V d1-7 and 15-21 every 28 days plus 100 mg E daily Dose level 3: 400 mg V d1-7 and 15-21 every 28 days plus 150 mg E daily
  Phase II:
  Dose level 3: 400 mg V d1-7 and 15-21 every 28 days plus 150 mg E daily
  Other Names: Zolinza® and Tarceva®

SUMMARY:
This is an open label, non-randomized, sequential, phase I/II trial in patients with stage IIIB or IV non-small cell lung cancer (NSCLC) with EGFR mutations after progression to Erlotinib. The study will have two parts. The first part (phase I) will be a dose finding (MTD) study to be implemented at three hospitals. The second part of the study (phase II) will asses the safety and efficacy of the combination. In this second part (phase II) patients will be treated with oral Erlotinib 150 mg P.O daily plus oral Vorinostat administered according to the results of the phase I. The study endpoints to be evaluated will include safety and response rate (RR) as primary endpoints and clinical benefit rate (CBR), time to progression, time to response, response duration and progression free survival as secondary endpoints. All the patients (phase I and II) will be treated until progression disease, unacceptable toxicity or withdrawal of the consent, and will be treated at the discretion of the principal investigator.

DETAILED DESCRIPTION:
SAMPLE:

Patients must have histologically-confirmed diagnosis of stage IIIB or IV NSCLC, with prior treatment with Erlotinib. In the phase I study the upper expected number of patients will be eighteen. In the phase II thirty two eligible patients will be included in the study. The enrollment period will be approximately 1.5 years. All patients will be treated with Erlotinib and Vorinostat regimen. Participating hospitals will be those of the Spanish Lung Cancer Group (SLCG).

For the phase I portion, there will be 3 sites: Dr. Noemi Reguart and Dr. Rafael Rosell, Institut Catala d'Oncologia, Hospital Germans Trias i Pujol, Badalona (Barcelona, Spain), Dr. Felip Cardenal, Institut Catalan d'Oncologia. Centre Sanitari i Universitari de Bellvitge (CSUB), Hospitalet de Llobregat (Barcelona, Spain) and Dr. Lola Isla, Hospital Clinico Lozano Blesa, (Zaragoza, Spain) For the phase II portion, 10 hospitals (adding 7 to the first 3) from the Spanish Lung Cancer Group (SLCG) will be involved. Hospitals will be included during phase I study.

OBJECTIVES AND HYPOTHESES Primary Phase I

(1) To determine the MTD of oral vorinostat in combination with erlotinib and to ensure that this treatment is sufficiently safe and tolerable to permit further study.

Phase II (1) To determine the percentage of patients free of progression at 12 weeks. Hypothesis: We considered that treatment was effective if we obtained a percentage of patients free of progression at 12 weeks higher than 60%.

Secondary

(1) To determine the CBR (clinical benefit rate), response rate, time to progression, time to response, response duration, and progression free survival in patients treated with vorinostat and erlotinib in combination.

Hypothesis: CBR should be of at least 25% and it will include stable disease for at least 3 months and objective RECIST response for at least 4 weeks.

Exploratory endpoints

Molecular analysis:

Main Objective: analysis of EGFR mutations (in exons 19, 20 and 21) in serum samples at baseline (before treatment), at three months of treatment and at the end of the treatment.

Secondary Objectives: retrospective analysis of molecular markers potentially related to drug sensitivity such as E-catherin protein expression, thioredoxin serum levels; Hsp70; methylation of 14-3-3r and CHFR.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed NSCLC
2. Diagnosis of advanced stage IIIB with pleural effusion or IV NSCLC
3. Previous disease progression after >= 3 months treatment with Erlotinib. Must tolerate erlotinib dose of 150 mg daily during the prior month.
4. Have demonstrated mutations at epidermal growth factor receptor (EGFR) at Exon 19 or Exon 21 (Exon 19 mutations characterized by in-frame deletions (747-750), and Exon 21 mutations resulting in L858R substitutions).
5. At least 18 years old.
6. Measurable disease as defined by the presence of at least one lesion that can be accurately measured in at least one dimension using RECIST guidelines.
7. At least 4 weeks from any prior major surgery or radiation therapy and have adequately recovered from the toxicities and/or complications
8. ECOG performance status 0 to 2
9. Adequate bone marrow function without the current use of colony stimulating factors.
10. Adequate coagulation function.
11. Adequate liver function
12. Adequate renal function
13. Non-sterilized premenopausal female, pregnancy test must be performed and patient must agree to use barrier methods of contraception. Male patients must agree to use an adequate method of contraception.
14. Available for periodic blood sample analyses, study related assessments 15.Patient has the ability to understand and willingness to sign the informed consent form.

16.Patient is able to read, understand, and complete the study questionnaires.

Exclusion Criteria:

1. Patient has been treated with any investigational agent for any indication within 4 weeks of study treatment.
2. Patient previously treated with Vorinostat or any other HDAC inhibitor for any indication in the previous 30 days.
3. Patient has history of hypersensitivity or intolerance to Erlotinib.
4. Patient has an active infection or has received intravenous antibiotic, antiviral or antifungal medications with 2 weeks
5. Patient with symptomatic central nervous system metastases with or without corticosteroids treatment.
6. Inability to take and/or tolerate oral medications.
7. Patient has known active hepatitis B or C infection,(HIV) HIV-related malignancy.
8. Pregnant or breastfeeding.
9. Patient with a history of gastrointestinal disease, surgery
10. Patient with uncontrolled undercurrent illness or circumstances that could limit compliance with the study.
11. History of malignancy except for inactive non-melanoma skin cancer and/or in situ carcinoma of the cervix, or other solid tumor treated curatively and without evidence of recurrence for at least 5 years prior to study enrollment.
12. Patient has had prescription or non-prescription drugs or other products known to influence CYP3A4 that cannot be discontinued prior to day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Moran, MD, Principal Investigator — Medical Oncology Service. Institut Catala d'Oncologia- ICO. Hospital Germans Trias i Pujol. Badalona - Barcelona (Spain); Dolores Isla, MD, Study Chair — Medical Oncology Service. Hospital Clinico Lozano Blesa. Zaragoza. Spain; Felip Cardenal, MD, Study Chair — Institut Catala d'Oncologia. Centre Sanitari i Universitari de Bellvitge (CSUB). Hospitalet de Llobregat (Barcelona). Spain; Bertomeu Massutti, MD, Study Chair — Medical Oncology Service. General Hospital. Alicante. Spain; Rafael Rosell, MD, Study Chair — Medical Oncology Service. Institut Catala d'Oncologia- ICO. Hospital Germans Trias i Pujol. Badalona - Barcelona (Spain); Noemi Reguart, MD, Study Chair — Medical Oncology Service. Hospital Clinic - Barcelona (Spain); Amelia Insa, MD, Principal Investigator — Medical Oncology Service. Hospital Clínico Universitario - Valencia (Spain); Cinta Pallarés, MD, Principal Investigator — Medical Oncology Service. Hospital de la Santa Creu i Sant Pau - Barcelona (Spain)
Locations (8):
- Spain (8):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Instituto Universitario Dexeus, Barcelona
  - Hospital Clinic, Barcelona
  - Institut Catalá d'Oncologia, Centre Sanitari i Universitari de Bellvitge (CSUB), Barcelona
  - Institut Catalá d'Oncología, Hospital Germans Trias i Pujol, Barcelona
  - Hospital La Paz, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clínico Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reguart N, Rosell R, Cardenal F, Cardona AF, Isla D, Palmero R, Moran T, Rolfo C, Pallares MC, Insa A, Carcereny E, Majem M, De Castro J, Queralt C, Molina MA, Taron M. Phase I/II trial of vorinostat (SAHA) and erlotinib for non-small cell lung cancer (NSCLC) patients with epidermal growth factor receptor (EGFR) mutations after erlotinib progression. Lung Cancer. 2014 May;84(2):161-7. doi: 10.1016/j.lungcan.2014.02.011. Epub 2014 Mar 2. PMID 24636848
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2007 and November 2010 the patients were enrolled in the phase I-II trial.
Pre-assignment Details: Screening details:
  Histologically confirmed NSCLC Diagnosis of advanced stage IIIB with pleural effusion or IV NSCLC Previous disease progression after >= 3 months treatment with Erlotinib. Must tolerate erlotinib dose of 150 mg daily during the prior month. Have demonstrated mutations at epidermal growth factor receptor (EGFR) at Exon 19 or Exon 21
Groups:
- Vorinostat Plus Erlotinib Phase II: Vorinostat plus Erlotinib
  Phase II:
  400 mg Vorinostat d1-7 and 15-21 every 28 days plus 150 mg Erlotinib daily per cycle
- Vorinostat Plus Erlotinib Phase I Level 1: Phase I:
  Dose level 1: 300 mg V d1-7 every 21 days plus 100 mg E daily If none of the patient experienced dose limiting toxicity, the next dose level was started.
- Vorinostat Plus Erlotinib Phase I Level 2: Dose level 2: 400 mg V d1-7 every 21 days plus 100 mg E daily Dose level 2b: 300 mg V d1-7 and 15-21 every 28 days plus 100 mg E daily
  If none of the patient experienced dose limiting toxicity, the next dose level was started.
- Vorinostat Plus Erlotinib Phase I Level 3: Dose level 3: 400 mg V d1-7 and 15-21 every 28 days plus 150 mg E daily
Period: Overall Study
Arm/Group | Vorinostat Plus Erlotinib Phase II | Vorinostat Plus Erlotinib Phase I Level 1 | Vorinostat Plus Erlotinib Phase I Level 2 | Vorinostat Plus Erlotinib Phase I Level 3
Started | 25 | 3 | 3 | 2
Completed | 25 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vorinostat Plus Erlotinib Phase II: Vorinostat plus erlotinib
  Phase II:
  Dose level 3: 400 mg V d1-7 and 15-21 every 28 days plus 150 mg E daily
- Vorinostat Plus Erlotinib Phase I: Drug: Vorinostat plus Erlotinib
  Phase I:
  Dose level 1: 300 mg V d1-7 every 21 days plus 100 mg E daily
- Vorinostat Plus Erlotinib Phase I Level 2: Drug: Vorinostat plus Erlotinib
  Phase I:
  Dose level 2: 400 mg V d1-7 every 21 days plus 100 mg E daily Dose level 2b: 300 mg V d1-7 and 15-21 every 28 days plus 100 mg E daily
- Vorinostat Plus Erlotinib Phase I Level 3: Drug: Vorinostat plus Erlotinib
  Phase I:
  Dose level 3: 400 mg V d1-7 and 15-21 every 28 days plus 150 mg E daily
- Total: Total of all reporting groups
Arm/Group | Vorinostat Plus Erlotinib Phase II | Vorinostat Plus Erlotinib Phase I | Vorinostat Plus Erlotinib Phase I Level 2 | Vorinostat Plus Erlotinib Phase I Level 3 | Total
Number analyzed (Participants) | 25 | 3 | 3 | 2 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.10) | 60 (9.93) | 54.67 (9.74) | 65 (12) | 60.12 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 1 | 1 | 1 | 19
  Male | 9 | 2 | 2 | 1 | 14
Region of Enrollment [Number; unit: participants]
  Spain | 25 | 3 | 3 | 2 | 33
ECOG [Number; unit: participants] — ECOG Performance Status Scale: It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability
  GRADES:
  ECOG 0: Fully active. ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours ECOG 4: Completely disabled ECOG 5: Dead
  participants
    ECOG 0 | 8 | 2 | 2 | 1 | 13
    ECOG 1 | 15 | 1 | 1 | 1 | 18
    ECOG 2 | 2 | 0 | 0 | 0 | 2
Smoking habits [Number; unit: participants]
  Current | 3 | 0 | 0 | 0 | 3
  Former > 5 years | 4 | 0 | 0 | 0 | 4
  Former 1-5 years | 1 | 0 | 0 | 0 | 1
  Former < 1 year | 1 | 0 | 0 | 0 | 1
  Never | 16 | 0 | 0 | 0 | 16
  Not recorded | 0 | 3 | 3 | 2 | 8
Stage [Number; unit: participants] — Staging is a classification where cancer is located, if or where it has spread and whether it's affecting other parts of the body.
  There are 5 stages for NSCLC:
  Stage 0:tumor hasn't grown into nearby normal lung tissues Stage I:small tumor that hasn't spread to any lymph nodes Stage II: medium tumor that hasn't spread to the nearby lymph nodes or N1 Stage III: cancer spread to the lymph nodes but haven't spread to other distant parts of the body Stage IV: cancer has spread to more than 1 area in the other lung, the fluid surrounding the lung or the heart, or distant parts of the body
  participants
    IIIB | 1 | 0 | 0 | 0 | 1
    IV | 24 | 3 | 3 | 2 | 32
Histology [Number; unit: participants]
  Adenocarcinoma | 21 | 3 | 3 | 2 | 29
  Squamous | 2 | 0 | 0 | 0 | 2
  Large cell | 2 | 0 | 0 | 0 | 2
Metastatic sites [Number; unit: participants]
  One | 5 | 0 | 0 | 0 | 5
  Two | 10 | 0 | 0 | 0 | 10
  Three or more | 10 | 0 | 0 | 0 | 10
  Not recorded | 0 | 3 | 3 | 2 | 8
EGFR tumor mutations [Number; unit: participants]
  Del 19 | 15 | 2 | 2 | 2 | 21
  L858R | 10 | 1 | 1 | 0 | 12
EGFR mutations blood [Number; unit: participants]
  Del 19 | 7 | 3 | 2 | 1 | 13
  L858R | 5 | 0 | 1 | 1 | 7
  Wild type | 6 | 0 | 0 | 0 | 6
  NE | 7 | 0 | 0 | 0 | 7
T790M blood [Number; unit: participants]
  Positive | 7 | 0 | 0 | 0 | 7
  Wild type | 11 | 0 | 0 | 0 | 11
  NE | 7 | 3 | 3 | 2 | 15
Median prior treatments [Number; unit: participants]
  One | 7 | 0 | 0 | 0 | 7
  Two | 4 | 0 | 0 | 0 | 4
  Three | 8 | 0 | 0 | 0 | 8
  Four or more | 6 | 0 | 0 | 0 | 6
  Not recorded | 0 | 3 | 3 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate at 12 Weeks
Description: Progression Free Survival was defined as time from first treatment until progression or death from any cause.
Time Frame: From date of first day of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 weeks
Population: Efficacy analysis PFSR12w population: all patients who have received at least one dose of study medication have been included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vorinostat Plus Erlotinib Phase II
Number analyzed (Participants) | 22
percentage of participants | 28 [18 to 37.2]

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Oral Vorinostat Phase I
Description: In the phase I, a classic 3 + 3 dose escalation method with 3 patients treated initially at each dose level was used. MTD was determined by testing on dose escalation cohorts: continuous full dose of erlotinib 150 mg orally (p.o.) in a daily administration(QD) and escalating doses of vorinostat p.o. at three dose levels:300 mg QD 7 days every 21 days, 400 mg QD 7 days every 21 days,and 400 mg QD, 7 days every other week. MTD reflects the highest dose of drug that did not cause a Dose-Limiting Toxicity (DLT) in less than or equal to 1 in 6 patients. DLTs were defined as any Vorinostat-related Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE 3.0) Grade 3 or 4 adverse events.
Time Frame: Up to 24 weeks for each dosing cohort
Population: Fourteen patients were treated with escalation doses of vorinostat.
Measure: Number; unit: mg
Groups:
- Vorinostat Plus Erlotinib Phase I: Vorinostat plus erlotinib
  Vorinostat plus Erlotinib: Phase I:
  Dose level 1: 300 mg V d1-7 every 21 days plus 100 mg E daily Dose level 2: 400 mg V d1-7 every 21 days plus 100 mg E daily Dose level 2b: 300 mg V d1-7 and 15-21 every 28 days plus 100 mg E daily Dose level 3: 400 mg V d1-7 and 15-21 every 28 days plus 150 mg E daily
Arm/Group | Vorinostat Plus Erlotinib Phase I
Number analyzed (Participants) | 14
mg | 400

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as time from study inclusion until death
Time Frame: From the date of study inclusion until end of follow up, up to 36 months.
Population: Efficacy analysis: all patients who have received at least one dose of study medication have been included.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Vorinostat Plus Erlotinib Phase II
Number analyzed (Participants) | 25
Month | 10.3 [2.4 to 18.1]

4. Secondary Outcome: Time to Progression
Description: The time to progression has been defined as the time that elapses, in months, since the patient begins study treatment until the patient progresses or dies from the disease, the first thing that occurs. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From the date of randomization until end of follow up, up to 36 months.
Population: Efficacy analysis: all patients who have received at least one dose of study medication have been included.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Vorinostat Plus Erlotinib Phase II
Number analyzed (Participants) | 25
Month | 1.8 [1.7 to 2]

ADVERSE EVENTS:
Time Frame: 37 months
Groups:
- Vorinostat Plus Erlotinib Phase I Dose Level 1: Dose level 1: 300 mg V d1-7 every 21 days plus 100 mg E daily If none of the patient experienced dose limiting toxicity, the next dose level was started.
- Vorinostat Plus Erlotinib Phase I Dose Level 2: Dose level 2: 400 mg V d1-7 every 21 days plus 100 mg E daily Dose level 2b: 300 mg V d1-7 and 15-21 every 28 days plus 100 mg E daily. If none of the patient experienced dose limiting toxicity, the next dose level was started.
- Vorinostat Plus Erlotinib Phase I Dose Level 3: Dose level 3: 400 mg V d1-7 and 15-21 every 28 days plus 150 mg E daily
Arm/Group | Vorinostat Plus Erlotinib Phase II | Vorinostat Plus Erlotinib Phase I Dose Level 1 | Vorinostat Plus Erlotinib Phase I Dose Level 2 | Vorinostat Plus Erlotinib Phase I Dose Level 3
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/3 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 16/25 | 0/3 | 1/3 | 2/2
Other Adverse Events (participants affected / at risk) | 22/25 | 3/3 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Vorinostat Plus Erlotinib Phase II (N=25) | Vorinostat Plus Erlotinib Phase I Dose Level 1 (N=3) | Vorinostat Plus Erlotinib Phase I Dose Level 2 (N=3) | Vorinostat Plus Erlotinib Phase I Dose Level 3 (N=2)
Fatigue (General disorders) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Pneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0 (0)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat Plus Erlotinib Phase II (N=25) | Vorinostat Plus Erlotinib Phase I Dose Level 1 (N=3) | Vorinostat Plus Erlotinib Phase I Dose Level 2 (N=3) | Vorinostat Plus Erlotinib Phase I Dose Level 3 (N=2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 20 (20) | 0 (0) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Ocular toxicity (Eye disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 16 (16) | 2 (2) | 1 (1) | 2 (2)
Asthenia (General disorders) | 10 (10) | 2 (2) | 1 (1) | 2 (2)
Anorexy (General disorders) | 9 (9) | 0 (0) | 2 (2) | 2 (2)
Fever (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 20 (20) | 2 (2) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 9 (9) | 0 (0) | 0 (0) | 2 (2)
Epigastralgia (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2)
Xerostomia (Gastrointestinal disorders) | 6 (6) | 2 (2) | 2 (2) | 2 (2)
Mucositis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Creatinine elevation (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 12 (12) | 1 (1) | 1 (1) | 2 (2)
Xeroderma (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was stopped prematurely because it did not meet the goal required for study continuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No